CLINICAL TRIAL: NCT01254175
Title: Phase 1 Study to Determine the Safety, Infectivity, Immunogenicity and Tolerability of 2 Doses of Live Attenuated Recombinant Cold-passaged (cp) 45 Human Parainfluenza Type 3 Virus Vaccine, rHPIV3cp45, Lot PIV3#102A, Delivered as Nose Drops to HPIV3-Seronegative Infants and Children 6 to 36 Months of Age, at a 6 Month Interval
Brief Title: Evaluating the Safety and Immunogenicity of a Human Parainfluenza Type 3 (HPIV3) Virus Vaccine in Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P1096; 11796 (Registry Identifier: DAIDS ES Registry Number); IMPAACT P1096
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Parainfluenza Virus 3, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rHPIV3cp45 Vaccine (Experimental): Participants will receive one dose of the rHPIV3cp45 vaccine at baseline and a second dose at Month 6.
  Interventions: Biological: rHPIV3cp45 Vaccine
- Placebo Vaccine (Placebo Comparator): Participants will receive one dose of the placebo vaccine at baseline and a second dose at Month 6.
  Interventions: Biological: Placebo Vaccine

INTERVENTIONS:
Biological: rHPIV3cp45 Vaccine — 10^5 TCID^50 of rHPIV3cp45 vaccine, delivered as nose drops
  Arms: rHPIV3cp45 Vaccine
Biological: Placebo Vaccine — Placebo vaccine, delivered as nose drops
  Arms: Placebo Vaccine

SUMMARY:
Human parainfluenza virus type 3 (HPIV3) is a major cause of pneumonia and other respiratory diseases in infants and children. This study will evaluate the safety and immune response of an HPIV3 vaccine in infants and young children.

DETAILED DESCRIPTION:
Human parainfluenza viruses can cause serious respiratory tract disease in infants and children under 5 years of age, and approximately 25% of children under 5 years of age have experienced a clinically significant parainfluenza virus infection. HPIV3, one of the four types of the parainfluenza virus, can cause pneumonia, bronchiolitis, croup, and bronchitis, and virtually all children have experienced primary HPIV3 infections by the time they are 3 to 4 years of age. In the United States, HPIV3 is responsible for approximately 11% of hospitalizations for respiratory diseases in children. Because HPIV3-associated lower respiratory illness typically occurs in the first year of life, the need exists for an HPIV3 vaccine that is safe and effective in infants. The purpose of this study is to evaluate the safety and immunogenicity of two doses of a live attenuated HPIV3 vaccine in infants and young children.

This study will enroll healthy, HPIV3 seronegative infants and children 6 months to 36 months of age. Participants will be randomly assigned to receive either the HPIV3 vaccine or a placebo vaccine. At a baseline study visit, all participants will undergo a medical history review, physical examination, vital sign measurements, and a nasal wash procedure. They will then receive their assigned vaccine in the form of nose drops. Participants will remain in the study clinic for 30 minutes after the vaccination for monitoring. Participants' parents will receive a thermometer and will record participants' temperature for 18 days after the vaccination. Study staff will call participants' parents on Days 1-18, 84, 112, and 140 to monitor participants' temperature and medical status. Study visits will occur 3, 6, 12, and 56 days after the vaccination, and participants will undergo similar tests and procedures as at the vaccination visit; a blood collection will also occur at Day 56. Six months after the first vaccination, all participants will return to the clinic and receive the second vaccination. All study procedures and study visits that followed the first vaccination will be repeated, and participants' last follow-up visit will occur 31 days after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian(s) of participants can demonstrate their understanding of the study (by taking a multiple choice questionnaire), sign the informed consent, and agree to vaccine administration following a detailed explanation of the study
* Seronegative for HPIV3, as defined by serum antibody titer hemagglutination inhibition (HAI) less than or equal to 1:8, as determined within 30 days prior to inoculation
* Medical history has been reviewed and a physical examination indicates that participant is in good health
* In the view of the site investigator, participant has received routine immunizations appropriate for age, administered at least 2 weeks prior to study entry (inactivated and subunit vaccines and rotavirus vaccine), or at least 4 weeks prior to study entry (live vaccines except rotavirus vaccine)
* Available for the entire study period and parent/guardian can be reached by telephone for post-inoculation contacts
* For children born to HIV-infected women, the child can be considered HIV-uninfected if he/she has either two negative polymerase chain reaction (PCR) tests with one collected at greater than 1 month of age and one collected at greater than 4 months of age, or two negative antibody tests
* If there is an immunocompromised child in the household who is less than 5 years of age, his/her last CD4 count must be greater than 15%

Exclusion Criteria:

* Known or suspected impairment of immunological functions, HIV infection, or currently (within the 30 days prior to study entry) receiving immunosuppressive therapy, including systemic corticosteroids (NOTE: Topical steroids, topical antibiotic, and topical antifungal medications are acceptable.)
* Bone marrow/solid organ transplant recipients
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with HPIV3 vaccine
* Previous serious vaccine-associated adverse event or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including reactive airway disease. People with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. People who wheezed once or received bronchodilator therapy once in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy in the 12 months before study entry may also be enrolled.
* Premature infants (born before 37 weeks gestation) if less than 12 months of age
* Members of a household which contains immunocompromised individuals (including, but not limited to, those with HIV-related immunodeficiency, defined as CD4 count less than 300 within the 6 months prior to study entry, or any household members who have received chemotherapy within the 12 months prior to study entry). More information on this criterion can be found in the protocol.
* Members of a household that contains infants less than 6 months of age
* Attends day care with infants less than 6 months of age and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. (Facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.)
* Participation in another investigational vaccine or drug trial within 30 days of receiving the investigational vaccine or until the final follow-up blood draw

Temporary Exclusion Criteria:

The following exclusion criteria are temporary or self-limiting conditions, and once resolved (after 24 hours and three normal measurements for fever) the infant may be enrolled, if otherwise eligible.

* Fever (rectal temperature of greater than or equal to 100.7 F), acute upper respiratory illness (including nasal congestion significant enough to interfere with successful vaccination), or acute otitis media
* Received any killed or subunit vaccine or rotavirus vaccine within the last 2 weeks; any live vaccine, except rotavirus, within the last 4 weeks; or gamma globulin (or other antibody products) within the past 3 months
* Received short-term systemic antibiotics for an acute illness within the 5 days prior to vaccination, or is currently receiving long-term prophylactic antibiotics (NOTE: Topical steroids, topical antibiotics, or topical antifungal preparations are permitted.)
* Received aspirin or aspirin-containing products within the 30 days prior to study entry
* Infants born at less than 37 weeks gestation will be deferred from participation until they are at least 12 months of age

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events that occur during the acute monitoring phase of the study | Measured at Days 0-18 after each vaccination
Proportion of participants that develop 4-fold or greater rises in hemagglutination inhibition (HAI) antibody titer following 2 doses of vaccine | Measured through 31 days after the second vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Coleen K. Cunningham, MD, Study Chair — Duke University
Locations (8):
- United States (7):
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Columbia IMPAACT CRS, New York, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - Seattle Children's Hospital CRS, Seattle, Washington
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Karron RA, Belshe RB, Wright PF, Thumar B, Burns B, Newman F, Cannon JC, Thompson J, Tsai T, Paschalis M, Wu SL, Mitcho Y, Hackell J, Murphy BR, Tatem JM. A live human parainfluenza type 3 virus vaccine is attenuated and immunogenic in young infants. Pediatr Infect Dis J. 2003 May;22(5):394-405. doi: 10.1097/01.inf.0000066244.31769.83. PMID 12792378
- [Background] Durbin AP, Karron RA. Progress in the development of respiratory syncytial virus and parainfluenza virus vaccines. Clin Infect Dis. 2003 Dec 15;37(12):1668-77. doi: 10.1086/379775. Epub 2003 Nov 20. PMID 14689350